CLINICAL TRIAL: NCT02655835
Title: Internet Mindfulness Meditation Intervention
Acronym: IMMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Helane Wahbeh, ND, MCR, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 10939
Record Dates: First submitted 2016-01-06; First posted 2016-01-14 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Stress
Keywords: mindfulness; meditation; internet

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet Mindfulness Meditation Intervention (Experimental): Six-week internet mindfulness meditation training program including handouts and daily guided meditations
  Interventions: Behavioral: Internet Mindfulness Meditation
- Access (Experimental): Written information handouts on mindfulness meditation and access to guided daily meditations
  Interventions: Behavioral: Access

INTERVENTIONS:
Behavioral: Internet Mindfulness Meditation
  Arms: Internet Mindfulness Meditation Intervention
Behavioral: Access
  Arms: Access

SUMMARY:
Phase 1 will follow 40 subjects and hopes to address whether or not IMMI can increase meditation practice as compared to another meditation program. The study will last six weeks for both the IMMI group (20 subjects) and the Access group (20 subjects). Access groups will receive learning materials and guided meditations, but the implementation will be self-paced. Participants in the IMMI group will receive weekly learning sessions and be required to practice meditation every day. IMMI group participants will also receive a weekly reminder call from a member of the study staff and have access to technical support in the event of trouble with the online program. All subjects will complete online self-report questionnaires that measure quality of life, self-efficacy, mood, sleep, mindfulness, and perceived stress at baseline and at the end of the six-week intervention. Subjects will also be given a questionnaire at the end of the study gauging their satisfaction with the mindfulness program they participated in.

Phase 2 will follow 80 subjects and hopes to address whether or not IMMI is acceptable to participants and demographic information about IMMI users. The study will be the same as noted above, but all subjects will be entered in the IMMI program.

Differences in recruitment rates, drop out, and patient satisfaction between the IMMI and Access groups will be analyzed. IMMI's ability to change meditation behavior (i.e. increasing time or frequency of meditation sessions), and improve quality of life will be examined as well.

DETAILED DESCRIPTION:
Participants will undergo the following: Week 0 - Telephone screening; Week 1 - Baseline Assessment; Week 2-Week 7 - Internet Mindfulness Meditation Intervention (or Access in Phase 1); Week 8 - Endpoint Assessment

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 80 years old
* Access to Computer and Internet
* Can hear and understand instructions
* Willing to accept randomization scheme and agrees to follow the study protocol

Exclusion Criteria:

* Significant acute medical illness that would decrease likelihood of study completion (self-report)
* Significant, untreated depression, as assessed by CESD-5 >20 during screening
* Current daily meditation practice (≥ 5 min/day daily for at least 30 days in the last 6 months. Past practice not exclusionary but will be recorded)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Enrollment rate | Week 0 - Screening
  Number of participants who are eligible and enroll in the study
Participant satisfaction | Week 8 - Endpoint assessment
  Client Satisfaction Questionnaire
Number of internet mindfulness meditation training sessions completed | Week 8 - Endpoint Assessment (after intervention is complete)
  There are a total of 6 internet training sessions, and participants are instructed to complete one per week (where Week 0 is screening, Week 1 is Baseline Assessment, Week 2 is Training 1, Week 3 is Training 2, Week 4 is Training 3, Week 5 is Training 4, Week 6 is Training 5, and Week 7 is Training 6) . At the time of the endpoint assessment (Week 8), the number of completed training sessions is tabulated.
Completion Rate | Week 8 - Endpoint assessment
  Number of participants who complete the endpoint assessment.

SECONDARY OUTCOMES:
Quality of Life SF-36 | Week 1 - Baseline assessment & Week 8 - Endpoint assessment
  Measured with Short-Form Health Survey (SF-36) self-report measure
Self-efficacy | Week 1 - Baseline assessment & Week 8 - Endpoint assessment
  Measured with General Perceived Self Efficacy (GPSE) self-report questionnaire
Mood | Week 1 - Baseline assessment & Week 8 - Endpoint assessment
  Measured with Center for Epidemiological Studies Depression Scale (CESD) self-report questionnaire
Sleep | Week 1 - Baseline assessment & Week 8 - Endpoint assessment
  Measured with Pittsburgh Sleep Quality Index (PSQI) self-report questionnaire
Mindfulness | Week 1 - Baseline assessment & Week 8 - Endpoint assessment
  Measured with Five Factor Mindfulness Questionnaire (FFMQ)
Perceived Stress | Week 1 - Baseline assessment & Week 8 - Endpoint assessment
  Measured with perceived stress scale (PSS)

CONTACTS AND LOCATIONS:
Overall Officials: Barry S Oken, MD, MS, Principal Investigator — Oregon Health and Science University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wahbeh H, Oken BS. Internet Mindfulness Meditation Intervention for the General Public: Pilot Randomized Controlled Trial. JMIR Ment Health. 2016 Aug 8;3(3):e37. doi: 10.2196/mental.5900. PMID 27502759